CLINICAL TRIAL: NCT00917670
Title: Ultrastructural Changes of Trabeculectomy Specimens in Patients With Uveitic Secondary Glaucoma
Status: Completed | Type: Observational
Sponsor: St. Franziskus Hospital (Other)
Collaborators: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Department of Ophthalmology at St. Franziskus Hospital
Other Study IDs: 2009-200-f-S-
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2010-07

CONDITIONS: Uveitis; Secondary Glaucoma
Keywords: trabecular meshwork; electron microscopy
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — trabeculectomy specimens including trabecular meshwork and Schlemms canal
Oversight: Data Monitoring Committee: No

SUMMARY:
Ultrastructural analysis of trabeculectomy specimens of patients with uveitic secondary glaucoma.

To evaluate morphological changes and to compare to primary open angle glaucoma patients.

ELIGIBILITY:
Inclusion Criteria:

* secondary uveitic glaucoma
* IOP > 24 mmhg with topical and/or systemic therapy
* need for surgical intervention to control IOP

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with uveitic secondary glaucoma in need of surgical intervention.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
morphological changes | after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anatomy II at University of Erlangen, Germany, Erlangen, Germany

REFERENCES:
- See also: Related Info — http://www.uveitis-zentrum.de